CLINICAL TRIAL: NCT05950568
Title: Efficacy of Quadratus Lumborum Block Type III Versus Type II Versus Transversus Abdominis Plane Block in Cesarean Section: A Randomized Controlled Multicenter Trial
Brief Title: Quadratus Lumborum Block Type III Versus Type II Versus Transversus Abdominis Plane Block in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The General Authority for Teaching Hospitals and Institutes (Network)
Responsible Party: Principal Investigator, Abeer Ali Elshabacy, Consultant of obstetrics and gynecology, The General Authority for Teaching Hospitals and Institutes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HB000132
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Cesarean Section; Quadratus Lumborum Block; Transversus Abdominis Plane Block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus lumborum block type II (Active Comparator): A 22 gauge needle was positioned between the erector spinae muscle in the thoracolumbar fascia's middle layer
  Interventions: Procedure: Quadratus lumborum block typen II
- Quadratus lumborum block type III (Active Comparator): A 22 gauge needle was positioned between the psoas and quadratus lumborum muscles at the anterior fascia lumbosacral
  Interventions: Procedure: Quadratus lumborum block III
- Transversus abdominis plane block (Active Comparator): A 22 gauge needle was positioned between the internal oblique and transversus abdominis muscles
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Quadratus lumborum block typen II — A 22 gauge needle was positioned between the quadratus lumborum muscle posterior border and the erector spinae muscle in the thoracolumbar fascia's middle layer
  Arms: Quadratus lumborum block type II
Procedure: Quadratus lumborum block III — A 22 gauge needle was positioned between the psoas and quadratus lumborum muscles at the anterior fascia lumbosacral
  Arms: Quadratus lumborum block type III
Procedure: Transversus abdominis plane block — A 22 gauge needle was positioned between the internal oblique and transversus abdominis muscles
  Arms: Transversus abdominis plane block

SUMMARY:
Compare the type III and type II quadratus lumborum block (QLB) to transversus abdominis plane block (TAPB) regarding efficacy in CS

DETAILED DESCRIPTION:
The transversus abdominis plane block (TAPB) is administered between the internal oblique muscle and the transversus abdominis muscle in the fascial plane, directly pointing to the somatic nerves T6-L1 that run in this plane. In addition, meta-analyses demonstrate that it is an effective analgesic for somatic pain and diminishes opiate intake. It has been reported that TAPB is an efficient analgesic approach following cesarean section .

The quadratus lumborum (QL) muscle block (QLB) is a fascial plane block as local anesthetic (LA) is introduced nearby to the QL muscle to numb the thoracolumbar nerves. QLB is categorized into four types according to drug administration location, I (lateral), II (posterior), III (anterior/transmuscular), and Intravenous, (intramuscular). QLB can effectively decrease both visceral and somatic pain by LA distribution to the thoracic paravertebral space (TPVS), as this block ensures effective pain control from the T7 to L1 dermatomes. QLB is one of the regional techniques that provides the greatest benefit in post-CS pain control, as it is progressively applied in obstetric anesthetic precise to improve analgesic results.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II
* aged 18 to 40 years old
* presenting for elective Cesarean section

Exclusion Criteria:

* body mass index (BMI) ≥40 kg/m2
* weight < 50kg
* height < 150 cm
* contraindications for the use of active labor, spinal anesthesia
* recent opiate intake
* hypersensitivity to any used medication
* substantial cardiovascular diseases
* renal diseases
* hepatic, diseases.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 60 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Total postoperative consumed pethidine | 24 hour postoperatively
  Numerical rating scales (NRS) score was evaluated at Post Anesthesia Care Unit (PACU), 2, 4, 6, 8, 12, 18, and 24 hours as as 0 is no pain and 10 is the worst pain imaginable. If the NRS score remained ≥ 4, we provided a bolus pethidine (0.5 mg/kg intravenous) and repeatable after 30 minutes if NRS remains≥ 4.

SECONDARY OUTCOMES:
Time of the first analgesic request | 24 hour postoperatively
  If the Numerical rating scales (NRS) score remained ≥ 4, we provided a bolus pethidine (0.5 mg/kg intravenous).
Patient satisfaction | 24 hour postoperatively
  The level of patient satisfaction was graded on a 5-point Likert scale as 0= extremely dissatisfied, 1= dissatisfied, 2= neither satisfied nor dissatisfied, 3= satisfied, 4= extremely satisfied
The degree of postoperative pain | 24 hour postoperatively
  Numerical rating scales (NRS ) score was evaluated at Post Anesthesia Care Unit (PACU), 2, 4, 6, 8, 12, 18, and 24 hours as as 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- The General Authority for Teaching Hospitals and Institutes, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author